CLINICAL TRIAL: NCT04660916
Title: Effects of Isotretinoin on the Morphology, Growth Rate, and Thickness of the Nail Plate
Brief Title: Effects of Isotretinoin on the Growth Rate and Thickness of the Nail Plate
Status: Completed | Type: Observational
Sponsor: Sinan Özçelik (Other)
Responsible Party: Sponsor-Investigator, Sinan Özçelik, Assistant Professor, Balikesir University
Organization: Balikesir University (Other)
Other Study IDs: 19AKD93
Record Dates: First submitted 2020-11-28; First posted 2020-12-09 (Actual); Last update posted 2020-12-09 (Actual); Status verified 2020-12

CONDITIONS: Isotretinoin; Nail Abnormality
Keywords: isotretinoin; nail growth rate; nail thickness; 13-cis-retinoic acid
MeSH Terms: conditions — Nails, Malformed | interventions — Isotretinoin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (2):
- isotretinoin: The patients aged 18-45 that were planned to begin treatment with isotretinoin for acne
  Interventions: Drug: Isotretinoin
- control: Healthy volunteers aged 18-45 without any diseases/drugs affecting the nail

INTERVENTIONS:
Drug: Isotretinoin — The effects of isotretinoin on morphology, growth rate, and thickness of the nail plate
  Other Names: Roaccutane; Zoretanin; D10BA01
  Groups: isotretinoin

SUMMARY:
The nail is an important skin appendage which can provide information about the person's overall health status in addition to having several important functions such as protection, tactile sensation, grasping. Many nail abnormalities which can have considerable psychological impact are side effects of drug administration. Retinoids have various effects on nails. Although isotretinoin as a retinoid has been associated with both decreased and increased nail growth, the great majority of such associations are not evidence-based. So, it was aimed to investigate the effects of isotretinoin on morphology, growth rate, and thickness of the nail plate.

DETAILED DESCRIPTION:
Isotretinoin has various side effects that affect many organ systems. Some side effects such as nail changes, which do not require treatment cessation, can limit the use of isotretinoin by impairing the patient's quality of life. Although it is known that isotretinoin has various effects on the nails, there is very limited data on effects of isotretinoin on the nails. Therefore, it was aimed to investigate the effect of isotretinoin on the morphology, growth rate, and thickness of the nail plate. The patients aged 18-45 that were planned to begin treatment with isotretinoin for acne in the outpatient clinic and a control group consisting of healthy volunteers are planned to be included in the study. A dermatological examination of skin and nails is conducted in all participants. Isotretinoin treatment at 0.5 mg/kg per day in 2 divided doses will be started to patients with acne. The length and thickness of nail plate are measured by digital caliper before isotretinoin treatment, and repeated during the control visits of the participants at 30 day intervals for 6 months. All the examination and measurements are carried out in both groups.

ELIGIBILITY:
Inclusion Criteria:

* The patients that were planned to begin treatment with isotretinoin for acne

Exclusion Criteria:

* Having known diseases (dermatological or systemic disorders) affecting the growth rate and thickness of nail plate
* Using systemic or topical drugs with known effects on nail
* Having traumatic nail abnormalities (onychotillomania, nail biting, habit-tic deformity)
* Having no visible lunula
* Describing any trauma (including cutting or filing nails) between the two measurements

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: All participants who are admitted to the outpatient clinic of our tertiary referral hospital were planned to include in the study.
Sampling Method: Non-Probability Sample
Enrollment: 70 (Actual)
Dates: Start 2019-10-22 (Actual); Primary Completion 2020-09-01 (Actual); Study Completion 2020-10-01 (Actual)

PRIMARY OUTCOMES:
The lengths and thicknesses of nail plate according to months in the isotretinoin group | 30 days
  These are the measures of monthly nail growth rates and thicknesses of nail plate. The lengths and thicknesses of nail plate are recorded in millimeters. Results are presented as mean or median according to whether they are normally distributed or not.
The lengths and thicknesses of nail plate according to months in the control group | 30 days
  These are the measures of monthly nail growth rates and thicknesses of nail plate. The lengths and thicknesses of nail plate are recorded in millimeters. Results are presented as mean or median according to whether they are normally distributed or not.
Comparison of nail growth rate according to groups | 30 days
  This is the comparison of monthly nail growth rates according to groups. The values of nail growth rates are recorded in millimeters per month.
Comparison of nail thickness according to groups | 30 days
  This is the comparison of monthly nail thickness according to groups. The values of nail thickness are recorded in millimeters.
The effect of group on the change in growth rate of nail plate by time | 30 days
  It is investigated using repeated measures analysis of variance
The effect of group on the change in thickness of nail plate by time | 30 days
  It is investigated using repeated measures analysis of variance
Changes in nail growth rates by time in the isotretinoin group | 30 days
  It is investigated using repeated measures analysis of variance
Changes in nail thickness by time in the isotretinoin group | 30 days
  It is investigated using repeated measures analysis of variance

CONTACTS AND LOCATIONS:
Overall Officials: Sinan Özçelik, MD, Principal Investigator — Balıkesir Üniversitesi
Locations (1):
- Balikesir University, Balıkesir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.